CLINICAL TRIAL: NCT00354432
Title: Randomized Study of Soy Protein and Effexor on Vasomotor Symptoms of Men With Prostate Cancer
Brief Title: Soy Protein/Effexor Hormone Therapy for Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped by the DSMB for lack of effect per interim stopping rule.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: REBAcccwfu97405; U10CA081851 (NIH)
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Hot Flashes; Prostate Cancer
Keywords: recurrent prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; hot flashes
MeSH Terms: conditions — Hot Flashes; Prostatic Neoplasms | interventions — Soybean Proteins; Isoflavones; Venlafaxine Hydrochloride; Caseins; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I - Placebo (Active Comparator): Patients receive oral placebo pill and oral placebo powder once daily.
  Interventions: Dietary Supplement: Placebo Powder; Drug: Placebo Pill
- Arm II - Soy (Active Comparator): Patients receive oral placebo pill and oral soy protein/isoflavones powder once daily.
  Interventions: Dietary Supplement: oral soy protein/isoflavones powder; Drug: Placebo Pill
- Arm III - Venlafaxine (Experimental): Patients receive oral Venlafaxine pill and placebo powder once daily.
  Interventions: Drug: Venlafaxine; Dietary Supplement: Placebo Powder
- Arm IV - Soy + Venlafaxine (Placebo Comparator): Patients receive oral Venlafaxine pill and soy protein/isoflavones powder once daily.
  Interventions: Dietary Supplement: oral soy protein/isoflavones powder; Drug: Venlafaxine

INTERVENTIONS:
Dietary Supplement: oral soy protein/isoflavones powder — Soy protein powder (20gm) orally 160 mg of total isoflavones isocaloric supplement of casein protein
  Other Names: Protein powder; Supplement powder soy and casein 20gm; Isoflavones; Isocaloric supplement; Casein protein
  Arms: Arm II - Soy; Arm IV - Soy + Venlafaxine
Drug: Venlafaxine — Patients receive oral venlafaxine 75mg.
  Other Names: Effexor XR; placebo
  Arms: Arm III - Venlafaxine; Arm IV - Soy + Venlafaxine
Dietary Supplement: Placebo Powder — Placebo powder (20gm casein protein) orally 0 mg of total isoflavones
  Other Names: Casein
  Arms: Arm I - Placebo; Arm III - Venlafaxine
Drug: Placebo Pill — Patients receive oral placebo pill.
  Other Names: Sugar Pill
  Arms: Arm I - Placebo; Arm II - Soy

SUMMARY:
RATIONALE: Soy protein/isoflavones and venlafaxine may help relieve hot flashes in patients receiving hormone therapy for prostate cancer. It is not yet known whether soy protein/isoflavones are more effective than venlafaxine when given together or with a placebo in treating hot flashes.

PURPOSE: This randomized phase III trial is studying soy protein/isoflavones and venlafaxine to compare how well they work when given together or with a placebo in treating hot flashes in patients receiving hormone therapy for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the effect of soy protein/isoflavones and venlafaxine on the hot flash symptom severity score in patients undergoing hormonal manipulation for treatment of prostate cancer.

Secondary

* Assess the effect of soy protein/isoflavones and venlafaxine on quality of life of these patients.
* Monitor and assess the participant drop out rate.

OUTLINE: This is a randomized, double-blind, multicenter study. Patients are stratified according to severity of disease (metastatic vs nonmetastatic) and baseline severity of hot flashes. Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive oral placebo pill and oral soy protein/isoflavones powder once daily.
* Arm II: Patients receive oral venlafaxine and oral placebo powder once daily.
* Arm III: Patients receive oral venlafaxine and oral soy protein/isoflavones powder once daily.
* Arm IV: Patients receive oral placebo pill and oral placebo powder once daily. Treatment in all arms continues for 12 weeks in the absence of disease progression or unacceptable toxicity. After 12 weeks of treatment, patients in arms I and III receive a tapered dose of oral venlafaxine once daily for 1 week.

Patients complete a vasomotor symptom diary once daily beginning 7 days before the initiation of study treatment and continuing until the completion of study treatment. Quality of life is assessed at baseline and at week 12.

PROJECTED ACCRUAL: A total of 176 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of prostate cancer, any stage Life expectancy of > nine months
* Prior or current androgen deprivation for treatment or control of prostate cancer to include:
* Bilateral Orchiectomy
* LHRH agonist (with or without antiandrogen therapy) ie: leuprolide (Lupron), goserelin (Zoladex), bicalutamide (Casodex), flutamide (Eulexin), or similar agents
* Chemotherapy
* Radiation (Patients may undergo concurrent radiation therapy to the prostate, prostate + seminal vesicles, and/or pelvis). Seed implants are allowed
* Participant report of hot flash frequency of an average of four or more per day, as defined by sweating, flushing, sensation of warmth, night sweats (Average of 28 per week)
* Hot flashes must be moderate or severe (See appendix A for hot flash definitions)
* Grade 2 (Moderate flashes) are warmer, produce obvious perspiration, and last 2 to 3 minutes
* Grade 3 (Severe flashes) causes profuse perspiration, generate intense heat, last longer and interfere with ongoing activity
* Age >21
* No allergies to soy or dairy products
* No current use of SSRIs, SNRI's, MAOIs, or Linezolide
* No uncontrolled hypertension (160/90) or greater than Class I American Heart Association functional capacity
* No history of mania, hypomania, bipolar disorder, or anorexia nervosa
* No history of seizures
* No history of hepatic dysfunction)
* Must have a telephone
* Signed protocol-specific Informed Consent
* Participants consuming soy foods or soy based supplements must continue on a stable regimen during study participation
* Patients should maintain same treatment and medications for prostate cancer throughout entire study.
* No change in treatment for 2 weeks prior to registration.
* Current use of medications and herbal supplements for hot flashes are allowed if on a stable regimen throughout the entire study. (Does not include anti-depressants)

Exclusion Criteria:

* Anticipated changes in prostate cancer treatment plan (i.e., hormonal manipulation, changes in chemotherapy)
* Concurrent antidepressant therapy
* History of intolerance to venlafaxine
* Recent (within 14 days) use of venlafaxine (Effexor XRTM), monoamine oxidase inhibitor, SSRI (selective serotonin reuptake inhibitor), or SNRI (selective norepinephrine reuptake inhibitor)
* History of seizure disorder

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-02-01 (Actual); Primary Completion 2010-08-01 (Actual); Study Completion 2010-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara Vitolins, DrPH, RD, Study Chair — Wake Forest University Health Sciences
Locations (20):
- United States (20):
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - MBCCOP - JHS Hospital of Cook County, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Heartland Research Consortium, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Southeastern Medical Oncology Center - Goldsboro, Goldsboro, North Carolina
  - Caldwell Memorial Hospital, Lenoir, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Wake Forest University CCOP Research Base, Winston-Salem, North Carolina
  - Cancer Centers of the Carolinas - Easley, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vitolins MZ, Griffin L, Tomlinson WV, Vuky J, Adams PT, Moose D, Frizzell B, Lesser GJ, Naughton M, Radford JE Jr, Shaw EG. Randomized trial to assess the impact of venlafaxine and soy protein on hot flashes and quality of life in men with prostate cancer. J Clin Oncol. 2013 Nov 10;31(32):4092-8. doi: 10.1200/JCO.2012.48.1432. Epub 2013 Sep 30. PMID 24081940

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm III - Venlafaxine: Patients receive oral venlafaxine pill and oral placebo powder once daily.
- Arm IV - Soy + Venlafaxin: Patients receive oral venlafaxine pill and oral soy protein/isoflavones powder once daily.
Period: Overall Study
Arm/Group | Arm I - Placebo | Arm II - Soy | Arm III - Venlafaxine | Arm IV - Soy + Venlafaxin
Started | 30 | 30 | 30 | 30
Completed | 24 | 22 | 20 | 20
Not Completed | 6 | 8 | 10 | 10
Not completed — Adverse Event | 3 | 1 | 5 | 5
Not completed — Off/Toxicity | 3 | 7 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Arm IV - Soy + Venlafaxine: Patients receive oral venlafaxine pill and oral soy protein/isoflavones powder once daily.
- Total: Total of all reporting groups
Arm/Group | Arm I - Placebo | Arm II - Soy | Arm III - Venlafaxine | Arm IV - Soy + Venlafaxine | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 12 | 11 | 43
  >=65 years | 19 | 21 | 18 | 19 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (8.8) | 71.0 (8.2) | 67.8 (9.9) | 67.5 (9.1) | 68.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 30 | 30 | 30 | 30 | 120
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 30 | 120

OUTCOME MEASURES:

1. Primary Outcome: Hot Flash Symptom Severity Score
Description: The primary objective of this randomized trial is to assess the effect of soy and Venlafaxine on the hot flash symptom severity score in men undergoing hormonal manipulation for treatment of prostate cancer. Hot flash severity will be quantitated using the symptom diary (as the sum of the number of hot flashes (any number greater than or equal to 0) times their severity (0=none, 1=mild, 2=moderate, 3=severe)). The primary end point is the 12 week hot flash score relative to the baseline value (i.e., 100*(12 week score)/baseline score). The range is 0 to infinity. Lower values represent a better outcome.
Time Frame: 12 weeks
Population: All randomized participants were analyzed in a repeated measures mixed model. This allowed inclusion of all study participants.
Measure: Least Squares Mean (Standard Error); unit: percent of baseline score
Arm/Group | Arm I - Placebo | Arm II - Soy | Arm III - Venlafaxine | Arm IV - Soy + Venlafaxine
Number analyzed (Participants) | 30 | 30 | 30 | 30
percent of baseline score | 52.3 (10.8) | 77.2 (11.6) | 68.9 (12.1) | 73.8 (11.9)
Statistical Analysis 1: Comparison: Arm I - Placebo vs Arm II - Soy vs Arm III - Venlafaxine vs Arm IV - Soy + Venlafaxine; The null hypothesis was that there was no difference in the hot flash severity score at 12 weeks; Test type: Superiority or Other; p = .3455, Mixed Models Analysis — This p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05; A mixed effects repeated measures analysis of variance was used with the baseline means constrained to be equal in the four groups

2. Secondary Outcome: Quality of Life
Description: Quality of life is quantified by the Functional Assessment of Cancer Therapy - Prostate questionnaire (FACT-P). The FACT-P consists of four general subscales (functional, emotional, social, and physical) consisting of a total of 27 questions as well as a Prostate specific subscale consisting of 12 questions. Each question is answered on a 0 to 4 scale. The FACT-P score ranges from 0 to 156; higher scores denote better quality of life.
Time Frame: 12 weeks
Population: Participants with baseline and 12 week quality of life data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I - Placebo | Arm II - Soy | Arm III - Venlafaxine | Arm IV - Soy + Venlafaxine
Number analyzed (Participants) | 21 | 21 | 18 | 17
units on a scale | 115.6 (2.4) | 121.5 (2.5) | 114.3 (2.7) | 117.7 (2.8)
Statistical Analysis 1: Comparison: Arm I - Placebo vs Arm II - Soy vs Arm III - Venlafaxine vs Arm IV - Soy + Venlafaxine; Null hypothesis was that there was no difference in quality of life between the four groups at 12 weeks; Test type: Superiority or Other; p = 0.2081, ANCOVA — This p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance was 0.05

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Arm I - Placebo | Arm II - Soy | Arm III - Venlafaxine | Arm IV - Soy + Venlafaxine
Serious Adverse Events (participants affected / at risk) | 4/30 | 5/27 | 5/29 | 5/28
Other Adverse Events (participants affected / at risk) | 28/30 | 23/27 | 29/29 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Placebo (N=30) | Arm II - Soy (N=27) | Arm III - Venlafaxine (N=29) | Arm IV - Soy + Venlafaxine (N=28)
Erectile Dysfunction (Reproductive system and breast disorders) | 2 (6) | 4 (13) | 2 (8) | 4 (13)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection - Rectum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood alteration - Agitation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood alteration- Anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstruction - Ureter (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (General disorders) | 2 (3) | 1 (1) | 1 (2) | 0 (0)
Pain - chest NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pain - joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular - other (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Placebo (N=30) | Arm II - Soy (N=27) | Arm III - Venlafaxine (N=29) | Arm IV - Soy + Venlafaxine (N=28)
Allergic Reaction/hypersensitivity including drug reaction (General disorders) | 1 (2) | 1 (4) | 2 (2) | 0 (0)
Anorexia (General disorders) | 4 (8) | 0 (0) | 3 (4) | 5 (12)
Confusion (Nervous system disorders) | 3 (3) | 0 (0) | 2 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 12 (23) | 5 (11) | 6 (15) | 10 (29)
Constitutional Symptioms - Nightmares (General disorders) | 2 (3) | 1 (1) | 2 (5) | 3 (9)
Diarrhea - without colostomy (Gastrointestinal disorders) | 6 (7) | 3 (3) | 5 (12) | 3 (7)
Distension/Bloating, Abdominal (Gastrointestinal disorders) | 6 (11) | 7 (14) | 10 (15) | 6 (12)
Dizziness (Ear and labyrinth disorders) | 6 (12) | 5 (11) | 7 (9) | 5 (9)
Dry Mouth (Gastrointestinal disorders) | 10 (28) | 6 (16) | 7 (10) | 7 (22)
Ejaculatory Dysfunction (Reproductive system and breast disorders) | 17 (58) | 11 (36) | 13 (39) | 12 (36)
Erectile Dysfunction (Reproductive system and breast disorders) | 17 (62) | 12 (42) | 13 (37) | 12 (32)
Fatigue (General disorders) | 18 (47) | 11 (36) | 18 (35) | 15 (36)
Flatulence (Gastrointestinal disorders) | 11 (22) | 9 (21) | 9 (17) | 11 (27)
Hypertension (Vascular disorders) | 4 (8) | 8 (17) | 4 (8) | 3 (8)
Insomnia (General disorders) | 15 (45) | 8 (20) | 11 (26) | 11 (26)
Mood Alteration - Agitation (Psychiatric disorders) | 3 (5) | 5 (10) | 7 (10) | 8 (12)
Mood Alteration - Anxiety (Psychiatric disorders) | 3 (10) | 4 (10) | 6 (11) | 3 (6)
Nausea (Gastrointestinal disorders) | 6 (9) | 3 (8) | 5 (6) | 8 (15)
Neurology - Nervousness (Nervous system disorders) | 3 (6) | 0 (0) | 1 (1) | 3 (7)
Neuropathy - Sensory (Nervous system disorders) | 2 (7) | 0 (0) | 1 (1) | 0 (0)
Pain - Other (General disorders) | 15 (38) | 13 (43) | 11 (32) | 8 (19)
Pain - Back (General disorders) | 0 (0) | 1 (4) | 2 (2) | 0 (0)
Pain - Extremity - Limb (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain - joint (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 0 (0) | 2 (3)
Petechiae/purpura - hemorrhage/bleeding into skin or mucosa (Skin and subcutaneous tissue disorders) | 1 (4) | 2 (6) | 0 (0) | 1 (3)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Somnolence (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (7)
Sweating - Diaphoresis (General disorders) | 20 (61) | 20 (64) | 24 (63) | 25 (74)
Urinary Frequency/Urgency (Renal and urinary disorders) | 2 (5) | 1 (4) | 2 (5) | 3 (8)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was stopped early by the DSMB due to a lack of effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes